CLINICAL TRIAL: NCT03913169
Title: Interprofessional Practice Education for Health Professional Students in Rural Communities
Brief Title: Interprofessional Practice Education for Health Professional Students
Acronym: HRSAIPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific Northwest University of Health Sciences (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, PNWU OSA, Executive Director of Interprofessional Education, Pacific Northwest University of Health Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2015-E-04
Record Dates: First submitted 2019-04-08; First posted 2019-04-12 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Interprofessional Relations
Keywords: Interprofessional Education; Medical Education; Interprofessional Practice; Doctor of Osteopathic Medicine; Physician Assistant

STUDY DESIGN:
Intervention Model Description: The intervention utilized in this project will involve a 2-year curriculum. The year one/pre-clinical curriculum will be presented to pre-clinical DO and PA students. The year two/clinical curriculum will be presented to third year Doctor of Osteopathic Medicine (DO) students and second year Physician Assistant (PA) students once clinic sites are identified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Students in Interprofessional Education Curriculum (Other): The interprofessional intervention for the students to be employed in this study will include five modalities in a scaffolded structure progressing from low- to high-fidelity experiences over a two-year period: (1) classroom didactic sessions; (2) simulation laboratory sessions; (3) standardized patient sessions; (4) community-based clinical case conferences; and, (5) community-based interprofessional rotations.
  Interventions: Other: Educational Implementation of Interprofessional Curriculum
- Patients Experience with Interprofessional Care (Other): For patients and their families, those who receive care from an Interprofessional team will receive the usual health care they normally receive at the participating clinics. In many cases patients already receive this care, but are unaware of it. Most of what occurs in Interprofessional practice happens outside of the patient encounter. For patients the process is generally invisible, but its affects are felt in terms of better communications with the patient. In this study, patients will be informed as usual about the presence of students as learners and will have the opportunity to decline student involvement in their care. The only difference for the patients and their families will be a request to fill out a survey form on paper indicating their perception of the experience in terms of quality of care and its potential impact on their access to care.
  Interventions: Other: Educational Implementation of Interprofessional Curriculum
- Clinician (Preceptor) Interprofessional Education Curriculum (Other): Clinicians will experience many of the same learning experiences as the students, but will differ in the level of education and its focus. Clinicians and faculty will be taught the concepts of Interprofessional education, the same as the students, but they will also be taught how to educate students using Interprofessional practices.
  Interventions: Other: Educational Implementation of Interprofessional Curriculum
- Faculty in Interprofessional Education Curriculum (Other): Doctor of Osteopathic Medicine and Physician Assistant Faculty will be taught the concepts of Interprofessional education, the same as the students, but they will also be taught how to educate students using Interprofessional practices.
  Interventions: Other: Educational Implementation of Interprofessional Curriculum

INTERVENTIONS:
Other: Educational Implementation of Interprofessional Curriculum — The intervention utilized in this project will involve a 2-year curriculum. The year one/pre-clinical curriculum will be presented to pre-clinical doctor of osteopathic medical students (DO) and physician assistant students (PA) students. The year two/clinical curriculum will be presented to third year DO students and second year PA students once clinic sites are identified.

SUMMARY:
The interprofessional practice & education curriculum for the students to be employed in this study will include five modalities in a scaffolded structure progressing from low- to high-fidelity experiences over a two-year period: (1) classroom didactic sessions; (2) simulation laboratory sessions; (3) standardized patient sessions; (4) community-based clinical case conferences; and, (5) community-based interprofessional rotations. Clinicians will experience many of the same learning experiences as the students, but will differ in the level of education and its focus. Clinicians and faculty will be taught the concepts of interprofessional practice & education, the same as the students, but they will also be taught how to educate students using interprofessional practice & education.

DETAILED DESCRIPTION:
The purpose of this prospective cohort study, which will utilize anonymous data, is to describe the impact of the interprofessional practice & education project in four categories:

1. Change in student knowledge, skill, and attitudes regarding interprofessional practice & education.
2. Student selection and entrance into primary care in rural settings and/or with underserved populations.
3. Patient and family members' perceptions of interprofessional practice & education encounters.
4. Clinicians' experiences with interprofessional practice & education and perceptions of it.

Research Questions:

1. How do students' knowledge, skill, and attitudes change regarding interprofessional practice & education as measured by pre/post electronic surveys?
2. What is the difference in the rate of entrance of graduates into primary care disciplines, settings that serve rural patients, and settings that serve underserved patients?
3. What are patients' and their families' perceptions of interprofessional practice & education encounters as measured by anonymous paper surveys.
4. What prior experiences and education do clinicians have with interprofessional practice & education?
5. How do clinicians' knowledge, skill, and attitudes change regarding interprofessional practice & education as measured by pre/post electronic surveys?

ELIGIBILITY:
Inclusion Criteria:

Students:

* Doctor of osteopathic medical students at Pacific Northwest University of Health Sciences
* Physician Assistant students at Heritage University
* Participants must also be over the legal age of consent

Clinicians (Preceptors):

* Affiliated Preceptors of Doctor of osteopathic medical students at Pacific Northwest University of Health Sciences
* Affiliated Preceptors of Physician Assistant students at Heritage University
* Participants must also be over the legal age of consent
* Interested in participating in this study by choosing whether they will complete the surveys.
* The five sites where this project will occur are already engaged in clinical case conferences and clinical rotations.

Patients:

* Patients included in this study must have a minimum of two conditions/diagnoses identified, such as diabetes, hypertension and coronary artery disease.
* These conditions could also include mental diagnoses, socioeconomic group, or other social determinants of health.
* Participants must also be over the legal age of consent.

Faculty:

* Faculty of the Doctor of osteopathic medical students at Pacific Northwest University of Health Sciences teaching specific concepts of Interprofessional Practice
* Faculty of the Physician Assistant students at Heritage University teaching specific concepts of Interprofessional Practice
* Participants must also be over the legal age of consent

Exclusion Criteria:

* Not enrolled as a student at Pacific Northwest University of Health Sciences Doctor of Osteopathic Medicine or Heritage University Physician Assistant Program
* Not an affiliated and approved clinical site of Pacific Northwest University of Health Sciences Doctor of Osteopathic Medicine or Heritage University Physician Assistant Program
* Patients unable to read or understand English at a 6th grade level

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1806 (Actual)
Dates: Start 2015-08-19 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Changes in Knowledge of Interprofessional Care and Practice Scores | Baseline and approximately 12-months from baseline
  Changes in Knowledge of Interprofessional Care and Practice Scores. The Knowledge of Interprofessional Care and Practice is designed to measure knowledge of under the umbrella of interprofessional collaborative practice over time. It is a 20 item quiz broken into 5 domains. Where incorrect answers "0" (to a very low knowledge) and correct answers "20" (to a very high knowledge).
Changes in Knowledge of Interprofessional Care and Practice Scores | Approximately 12-months to 24-months from baseline
  Changes in Knowledge of Interprofessional Care and Practice Scores. The Knowledge of Interprofessional Care and Practice is designed to measure knowledge of under the umbrella of interprofessional collaborative practice over time. It is a 20 item quiz broken into 5 domains. Where incorrect answers "0" (to a very low knowledge) and correct answers "20" (to a very high knowledge).
Changes in Knowledge of Interprofessional Care and Practice Scores | Episodic from Baseline to 24-months from baseline
  Changes in Knowledge of Interprofessional Care and Practice Scores. The Knowledge of Interprofessional Care and Practice is designed to measure knowledge of under the umbrella of interprofessional collaborative practice over time. It is a 20 item quiz broken into 5 domains. Where incorrect answers "0" (to a very low knowledge) and correct answers "20" (to a very high knowledge).
Changes in Interprofessional Learning Readiness Scale Scores | Baseline and approximately 12-months from baseline
  Changes in Interprofessional Learning Readiness Scale Scores. Interprofessional Learning Readiness Scale is designed to assess learning readiness/attitudes of health sciences students towards interprofessional teamwork and education perceptions of interprofessional collaboration Self-report (e.g., survey, questionnaire, self-rating), 18-item, 6-point likert-type scale ranging from strongly agree (6) to strongly disagree (1). A higher number indicating a stronger readiness versus a lower score.
Changes in Interprofessional Learning Readiness Scale Scores | Approximately 12-months to 24-months from baseline
  Changes in Interprofessional Learning Readiness Scale Scores. Interprofessional Learning Readiness Scale is designed to assess learning readiness/attitudes of health sciences students towards interprofessional teamwork and education perceptions of interprofessional collaboration Self-report (e.g., survey, questionnaire, self-rating), 18-item, 6-point likert-type scale ranging from strongly agree (6) to strongly disagree (1). A higher number indicating a stronger readiness versus a lower score.
Changes in Interprofessional Learning Readiness Scale Scores | Episodic from Baseline to 24-months from baseline
  Changes in Interprofessional Learning Readiness Scale Scores. Interprofessional Learning Readiness Scale is designed to assess learning readiness/attitudes of health sciences students towards interprofessional teamwork and education perceptions of interprofessional collaboration Self-report (e.g., survey, questionnaire, self-rating), 18-item, 6-point likert-type scale ranging from strongly agree (6) to strongly disagree (1). A higher number indicating a stronger readiness versus a lower score.
Changes in Team Performance Observation Tool Ratings | Baseline and approximately 12-months from baseline
  Changes in Team Performance Observation Tool Ratings. The Performance Observation Tool (TPOT) is a TeamSTEPPS®curriculum instrument that can be utilized to evaluate the effectiveness of team performance. It is a 5 domain, 23 item rating for the team. Rating Scale: 1 = Very Poor, 2 = Poor, 3 = Acceptable, 4 = Good, and 5 = Excellent. Where total ratings of "23" indicate low team performance and "115" indicate high team performance.
Changes in Team Performance Observation Tool Ratings | Approximately 12-months to 24-months from baseline
  Changes in Team Performance Observation Tool Ratings. The Performance Observation Tool (TPOT) is a TeamSTEPPS®curriculum instrument that can be utilized to evaluate the effectiveness of team performance. It is a 5 domain, 23 item rating for the team. Rating Scale: 1 = Very Poor, 2 = Poor, 3 = Acceptable, 4 = Good, and 5 = Excellent. Where total ratings of "23" indicate low team performance and "115" indicate high team performance.
Changes in Team Performance Observation Tool Ratings | Episodic during Baseline to Throughout 24-months
  Changes in Team Performance Observation Tool Ratings. The Performance Observation Tool (TPOT) is a TeamSTEPPS®curriculum instrument that can be utilized to evaluate the effectiveness of team performance. It is a 5 domain, 23 item rating for the team. Rating Scale: 1 = Very Poor, 2 = Poor, 3 = Acceptable, 4 = Good, and 5 = Excellent. Where total ratings of "23" indicate low team performance and "115" indicate high team performance.
Total Scores of Patient Perceived Quality of Care | Episodic from Baseline to 24-months from baseline
  The Patient Perceived Quality of Care satisfaction of the care the patient received with the collaborative and communicative aspects of care teams. The satisfaction is determined by this 7-item rating system of Yes- 3; Partly -2; No - 1; and Does not Apply - 0. Where total ratings of "0" indicate low perceived quality of care and "21" indicate high perceived quality of care.
Changes in Perception of Interprofessional Collaboration Model Questionnaire. | Baseline and approximately 12-months from baseline
  The Perception of Interprofessional Collaboration Model Questionnaire is designed to assess perceptions of interprofessional collaboration on the individual, group, and organizational levels for professionals in the domain of mental health care for children and adolescents. Self-report (e.g., survey, questionnaire, self-rating), 12 constructs 48-item, 7-point Likert-type scale ranging from strongly agree (1) to strongly disagree (7).
Changes in Perception of Interprofessional Collaboration Model Questionnaire. | Approximately 12-months to 24-months from baseline
  The Perception of Interprofessional Collaboration Model Questionnaire is designed to assess perceptions of interprofessional collaboration on the individual, group, and organizational levels for professionals in the domain of mental health care for children and adolescents. Self-report (e.g., survey, questionnaire, self-rating), 12 constructs 48-item, 7-point Likert-type scale ranging from strongly agree (1) to strongly disagree (7).
Changes in Perception of Interprofessional Collaboration Model Questionnaire. | Episodic from Baseline to 24-months from baseline
  The Perception of Interprofessional Collaboration Model Questionnaire is designed to assess perceptions of interprofessional collaboration on the individual, group, and organizational levels for professionals in the domain of mental health care for children and adolescents. Self-report (e.g., survey, questionnaire, self-rating), 12 constructs 48-item, 7-point Likert-type scale ranging from strongly agree (1) to strongly disagree (7).

CONTACTS AND LOCATIONS:
Overall Officials: Keith Monosky, PhD, Principal Investigator — Pacific Northwest University of Health Sciences
Locations (2):
- United States (2):
  - Heritage University, Toppenish, Washington
  - Pacific northwest university of health sciences, Yakima, Washington

IPD SHARING:
Plan to Share IPD: No